CLINICAL TRIAL: NCT06572241
Title: Quality of Labour Epidural Analgesia With Intrathecal Morphine as a Component of Combined Spinal Epidural: a Double-blinded Randomized Control Trial
Brief Title: Quality of Labour Epidural Analgesia With Intrathecal Morphine as a Component of Combined Spinal Epidural
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-06
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Labor Pain
Keywords: combined spinal epidural; CSE; intrathecal morphine
MeSH Terms: conditions — Labor Pain | interventions — Morphine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine (Active Comparator): 0.6 ml of 0.25% bupivacaine, fentanyl 10 mcg with morphine 100 mcg (total volume 1 ml) as intrathecal component of combined spinal epidural (CSE).
  Interventions: Drug: Intrathecal morphine
- Placebo (Placebo Comparator): 0.6 ml of 0.25% bupivacaine, fentanyl 10 mcg with normal saline 0.2 ml (total volume 1 ml) as intrathecal component of combined spinal epidural (CSE).
  Interventions: Other: Saline solution (placebo)

INTERVENTIONS:
Drug: Intrathecal morphine — morphine 100 mcg, included in the intrathecal component of combined spinal epidural (CSE).
  Other Names: Morphine
  Arms: Morphine
Other: Saline solution (placebo) — normal saline 0.2 ml added to the intrathecal component of combined spinal epidural (CSE).
  Other Names: saline
  Arms: Placebo

SUMMARY:
Neuraxial analgesia has shown to be the gold standard for effective labor pain relief, offering numerous benefits including enhanced pain control and maternal satisfaction. The methods to achieve neuraxial analgesia include lumbar epidural (LE), and combined spinal epidural (CSE). While LE may not consistently provide optimal pain relief, leading to frequent maternal requests for supplemental analgesics, CSE presents a promising advancement. This is due to the rapid onset of pain relief from intrathecal components, complemented by the longer-lasting effects of epidural medications. Intrathecal drugs have demonstrated the ability to offer more symmetrical blockades compared to epidurally administered medications. Nonetheless, some clinicians remain cautious about CSE due to the potential for increased pain when transitioning from spinal to less effective epidural analgesia. Long-acting opioids like morphine in the intrathecal space may mitigate this problem by providing transitional analgesia to the laboring parturient.

The primary aim of this randomized controlled trial is to provide evidence of whether the addition of 100 mcg of morphine in the intrathecal (spinal) component of CSE reduces the rate of breakthrough pain during labor.

DETAILED DESCRIPTION:
The addition of morphine to a combination of bupivacaine and lipophilic opioids (fentanyl) for the spinal component of CSE for labor analgesia has been shown to increase the duration of analgesia. A meta-analysis by Al-Kazwini and coworkers suggests a possible beneficial prolonging effect of adding morphine to spinal analgesia, however, the authors concluded that more adequately powered randomized controlled trials (RCTs) are required to determine the benefits and harms of intrathecal morphine (ITM).

This prolonged duration of action of ITM may reduce the need for frequent top-ups, which could alleviate nursing and anesthesiologist workload and enhance maternal satisfaction. An RCT conducted by Vasudevan and coworkers has concluded that the addition of 100 mcg ITM along with bupivacaine and fentanyl reduced the incidence of breakthrough pain in labor. Another dose-finding study comparing 50 and 100 mcg of ITM as a component of CSE labor analgesia concluded that 100 mcg of ITM significantly lowers the local anesthetic consumption and shorter duration of the first stage of labor without any significant difference in adverse effects. The RCT by Vasudevan et al. had a small sample size, enrolled mixed parity patients, and utilized continuous infusion for labor analgesia maintenance.

Hence, the investigators plan to conduct adequately powered RCT enrolling only primigravidae patients, which tend to have more prolonged labor than multiparous and programmed intermittent epidural bolus (PIEB) with patient-controlled epidural analgesia (PCEA) will be used, which is a more contemporary labor maintenance technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) term primiparous (≥37 weeks) patients with live singleton pregnancy
* Patients who request labour analgesia and do not have any contraindications for neuraxial analgesia.
* Less than or equal to 6 cm cervical dilation during the last vaginal examination.

Exclusion Criteria:

* Patients who are expected to be discharged within 24 hours of delivery.
* Patients with chronic pain conditions, opioid use disorder, pre-gestational diabetes, obstructive sleep apnea, morbid obesity (BMI >40 kg/m2), or fetal abnormalities.
* Patients who have intramuscular morphine within 12 hours or fentanyl >200 mcg in the preceding 4 hours.
* Participants will be excluded from further analysis in case of spinal analgesic failure
* Participants will be excluded from further analysis if labour lasts less than 2 hours

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 182 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Presence of breakthrough pain: questionnaire | 24 hours
  The rate of breakthrough pain is defined as the ratio of the number of episodes of breakthrough pain during labour analgesia and the duration of epidural analgesia. An episode of breakthrough pain during labour analgesia was defined as subjective discomfort due to pain or pressure increasing during a contraction (rated as NRS ≥3/10), which was successfully treated with the manual administration of supplemental medications.

SECONDARY OUTCOMES:
Time to first episode of breakthrough pain in minutes | 24 hours
  The amount of time in minutes to the first recorded episode of breakthrough pain, defined as subjective discomfort due to pain or pressure increasing during a contraction (rated as NRS ≥3/10), which was successfully treated with the manual administration of supplemental medications.
Epidural medication consumption (milliliters) | 24 hours
  The overall consumption of epidural medication throughout labour, in milliliters.
Epidural pump settings: questionnaire | 24 hours
  Any adjustments made to the programmed intermittent bolus settings of the epidural pump will be recorded.
Presence of fetal heart rate anomalies: questionnaire | 24 hours
  The presence of any fetal heart rate anomalies will be recorded
Presence of Cesarean delivery: questionnaire | 24 hours
  The presence of Cesarean delivery will be recorded
Analgesic consumption post-delivery: questionnaire | 24 hours
  Presence of analgesic consumption post-delivery will be recorded.
Presence of pruritis: questionnaire | 24 hours
  The presence of pruritis (yes or no) will be recorded.
Presence of nausea: questionnaire | 24 hours
  The presence of nausea(yes or no) will be recorded.
Presence of vomiting: questionnaire | 24 hours
  The presence of vomiting(yes or no) will be recorded.
Presence of sedation: questionnaire | 24 hours
  The presence of sedation(yes or no) will be recorded.
Presence of respiratory depression: questionnaire | 24 hours
  The presence of respiratory depression(yes or no) will be recorded.
Apgar score at 1 minute | 1 minute
  Apgar score recorded by the respiratory therapist, nurse or midwife at 1 minute of life.
Apgar score at 5 minutes | 5 minutes
  Apgar score recorded by the respiratory therapist, nurse or midwife at 5 minutes of life.
Umbilical artery pH | 24 hours
  Lab results for umbilical artery pH
Umbilical vein pH | 24 hours
  Lab results for umbilical vein pH
Satisfaction: questionnaire | 24 hours
  Post-delivery, patients will be asked how satisfied they were with their labour analgesia from 0-10, where 0 is no pain and 10 is the worst pain imaginable.
Obstetric Quality of Recovery-10 (ObsQoR-10) score 24 hours | 24 hours
  ObsQoR-10 score at 24 hours. There are 10 questions, and the results are tabulated out of 100. The higher the overall score out of 100, the better quality of recovery a patient is experiencing.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Siddiqui, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No